CLINICAL TRIAL: NCT07133191
Title: Single-center, Double-blind Trial to Assess the Pharmacokinetics, the Pharmacodynamics, and the Tolerability of a Single 16 mg Dose of Selatogrel (ACT-246475) in Healthy Japanese and Caucasian Participants
Brief Title: A Trial to Compare What the Body Does to Selatogrel and the Effect of Selatogrel in Japanese and Caucasian Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-076-110
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Selatogrel (Experimental): Study treatment is administered in the morning as a subcutaneous single dose.
  Interventions: Combination Product: Selatogrel
- Placebo (Placebo Comparator): Study treatment is administered in the morning as a subcutaneous single dose.
  Interventions: Combination Product: Matching placebo

INTERVENTIONS:
Combination Product: Selatogrel — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration.
  A single dose of 16 mg selatogrel will be administered as a liquid formulation from a sealed prefilled syringe in an autoinjector forming an integral ready-to-use, single-dose drug delivery system.
  Other Names: ACT-246475
  Arms: Selatogrel
Combination Product: Matching placebo — A single dose of placebo will be administered as a liquid formulation from a sealed prefilled syringe in an autoinjector forming an integral ready-to-use, single-dose drug delivery system.
  Arms: Placebo

SUMMARY:
This study is for research purposes only and is not intended to treat any medical condition. The purpose of this study is to evaluate the pharmacokinetics (PK), pharmacodynamics (PD), and tolerability of selatogrel following a single dose in healthy Japanese and Caucasian participants. Pharmacokinetics is the study of the absorption and breakdown of the study drug in the body. Pharmacodynamics is the study of the effect of the study drug on the body. There will be 2 groups in the study: 16 Japanese participants in one group and 16 Caucasian participants in the other group.

The duration of participation in this study is approximately 70 days from screening to the end of follow-up. A screening visit is required within 28 days prior to the start of the study to determine whether the volunteer qualifies and is willing to participate in this research study. This study requires in-patient stay in the research clinic of 3 or 4 days (2 or 3 nights), an end-of-trial (EOT) examination at least 36 hours after study drug administration, and a post-trial safety follow-up telephone call or site visit 30-40 days after the EOT examination.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent form in a language understandable to the participants prior to any trial-mandated procedure.
* Participant must be of either Caucasian (with European, North African, Middle Eastern origins) or Japanese ethnicity.
* Body mass index (BMI) of 18.0 to 28.0 kg/m2 (inclusive) at Screening.
* Systolic blood pressure 90-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on the dominant arm, after 5 min in the supine position at Screening.
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, measured after 5 min in the supine position at Screening.
* Clinical chemistry test results not deviating from the normal range to a clinically relevant extent at Screening.
* Hematology and coagulation test results not deviating from the normal range to a clinically relevant extent at Screening and on admission.
* Negative results from urine drug screen and alcohol breath test at Screening and on admission.
* Ability to communicate well with the investigator, in a language understandable to the participant, and to understand and comply with the requirements of the trial.
* For participants of childbearing potential: Negative results from serum pregnancy test at Screening and urine pregnancy test on admission. They must consistently and correctly use (from Screening, during the entire trial, and for at least 30 days after trial intervention injection) an acceptable method of contraception, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must be initiated at least 1 month before trial intervention administration.

Main Exclusion Criteria:

* Previous exposure to selatogrel.
* Pregnant or lactating participant.
* Known hypersensitivity to P2Y12 receptor antagonists or to excipients used in any of the formulations.
* Family or personal history of prolonged bleeding (e.g., after surgical intervention) or bleeding disorders (e.g., thrombocytopenia, clotting disturbances), intracranial vascular diseases, stroke, transient ischemic attack, reasonable suspicion of vascular malformations, peptic ulcers.
* Platelet count < 120 × 109 L-1 at Screening or on admission.
* Any known platelet disorder (e.g., Glanzmann thrombo-asthenia, von Willebrand disease, platelet release defect).
* Previous treatment with acetylsalicylate, non-steroidal anti-inflammatory drugs, P2Y12 receptor antagonists, or any medication with blood-thinning activity (i.e., injectable or oral anticoagulants) within 3 weeks prior to trial intervention administration.
* Treatment with another investigational small-molecule drug within 3 months or 5 × half-life (t1/2, whichever is longer) or with an investigational antibody treatment within 6 months prior to Screening, or participation in more than 4 investigational drug trials within 1 year prior to Screening.
* Excessive caffeine consumption from trial drug administration to EOT, defined as ≥ 800 mg per day at Screening.
* Nicotine use within 3 months prior Screening and inability to refrain from nicotine intake from Screening until EOT.
* History or clinical evidence of alcoholism or drug abuse within 3 years prior to Screening.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) with the exception of contraceptives for participants of childbearing potential within 2 weeks or 5 × t1/2 (whichever is longer) prior to study drug administration.
* History of major medical or surgical disorders, which in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed).
* History of asthma.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Legal incapacity or limited legal capacity or vulnerability (e.g., kept in detention) at Screening.
* Known hypersensitivity or allergy to natural rubber latex.
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the trial.
* Participant is the investigator or any delegate, research assistant, pharmacist, trial coordinator, other staff from trial site or the sponsor directly involved in the conduct of the trial or their relatives.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) | Up to 36 hours post-dose
  The plasma selatogrel PK parameters will be derived by non compartmental analysis of the concentration-time profiles
Area under the plasma concentration-time curve from zero to infinity (AUC0-infinity) | Up to 36 hours post-dose
  The plasma selatogrel PK parameters will be derived by non compartmental analysis of the concentration-time profiles
Maximum plasma concentration (Cmax) | Up to 36 hours post-dose
  The measured individual plasma concentrations of selatogrel will be used to directly obtain Cmax
Time to reach maximum plasma concentration (tmax) | Up to 36 hours post-dose
  The measured individual plasma concentrations of selatogrel will be used to directly obtain tmax
Terminal half-life (t1/2) | Up to 36 hours post-dose
  The plasma selatogrel PK parameters will be derived by non compartmental analysis of the concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- CenExel ACT (Anaheim Clinical Trials), Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No